#### MOD00003127 FSU IRB Approved 8 February 2023 

### **Permission to Take Part in a Human Research Study**

# Title of research study: Text Based Digital Interventions Prompting Enjoyable and Healthy Behaviors

Investigator: Greg Hajcak, Ph.D.

**Key Information:** We invite you to take part in an online research study.

First, we want you to know that:

Taking part in research is entirely voluntary.

You may choose not to take part, or you may withdraw from the study at any time. In either case, you will not lose any benefits to which you are otherwise entitled.

You may receive no benefit from taking part. The research may give us knowledge that may help people in the future.

Second, some people have personal, religious or ethical beliefs that may limit the kinds of research procedures they would want to receive. If you have such beliefs, please discuss them with the research team before you agree to the study.

Now we will describe this research study. Before you decide to take part, please take as much time as you need to ask any questions and discuss this study with anyone on the FSU research team (i.e., over the phone or email), or with family, friends or your personal physician or other professional.

### Why am I being invited to take part in a research study?

We invite you to take part in this research study because of your responses related to items of current depressive symptoms on our study screening.

### What should I know about a research study?

- This study will take place completely online
- Whether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.

## Why is this research being done?

This study is being conducted by Greg Hajcak, Ph.D., Psychology Department.

The purpose of the study is: to examine the effectiveness of one-month of text message reminders in reducing depressive symptoms. Engaging in both healthy self-care behaviors and enjoyable activities

### MOD00003127 FSU IRB Approved Page 2 of 5y 2023

### Permission to Take Part in a Human Research Study

may help reduce depressive symptoms—and the current study is designed to test whether text reminders to engage healthy self-care or enjoyable activities reduce depressive symptoms.

### How long will the research last and what will I need to do?

We expect that you will be in this research study for one month. You will first be asked to take a baseline survey lasting approximately one hour. Over the next four weeks, you may be sent daily reminders and brief checklists to fill out. You will also have a short weekly questionnaire to complete asking about your mood. At the end of the month, you will again complete a one-hour survey.

More detailed information about the study procedures can be found under "What happens if I say yes, I want to be in this research?"

### Is there any way being in this study could be bad for me?

The study has the following risks: discomfort in describing your thoughts and behaviors. Because this is a research study, there may be additional risks that we cannot identify at this time. More detailed information about the risks of this study can be found under "Is there any way being in this study could be bad for me? (Detailed Risks)"

#### Will being in this study help me anyway?

The benefits to study participation are: There is no direct benefit as a result of being in this study. Potential benefits include contributing to research that will help us understand the feasibility and effectiveness of programs that prompt people to engage in healthy behaviors.

#### What happens if I do not want to be in this research?

Participation in research is completely voluntary. You can decide to participate or not to participate.

#### MOD00003127 FSU IRB Approved Reprintly 2023 

### Permission to Take Part in a Human Research Study

**<u>Detailed Information:</u>** The following is more detailed information about this study in addition to the information listed above.

#### Who can I talk to?

If you have questions, concerns, or complaints, or think the research has hurt you, talk to the research team at hajcakip@gmail.com or at 850-320-7087.

This research has been reviewed and approved by an Institutional Review Board ("IRB"). You may talk to them at 850-644-7900 or humansubjects@fsu.edu if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research subject.
- You want to get information or provide input about this research.

# How many people will be studied?

We expect that about 150 participants will be in this research study.

# What happens if I say yes, I want to be in this research?

This study will be conducted completely online. At the start of the study, you will randomly be assigned to one of three conditions. One group of people will receive text reminders regarding enjoyable activities, the other will receive text reminders about healthy self-care behaviors, and the last will not receive any text reminds. Neither you nor the researcher will choose what condition you are assigned to. Regardless of which condition you are randomly assigned to, you will be able to complete the other condition at the end of the study if you would like; however, you will not be compensated if you opt to do that. In all conditions: you will complete an introduction video about your assigned intervention, followed by a pre-intervention survey, after which you will report on your desired enjoyable activities.

If you are in the enjoyable activities condition, you will receive daily reminders to do the activities you've selected from the list, as well as a checklist at the beginning of each day where you will report how frequently you have completed any of your chosen five activities from the previous day. You will also have a short weekly questionnaire to complete asking about your overall mood for that week.

If you are in the healthy self-care behaviors condition, you will be prompted to complete activities such as drinking enough water, going to bed early, reminders about good hygiene, and eating well-balanced meals. Daily text reminders will be sent about these healthy self-care activities. You will receive a checklist at the beginning of each day where you will report about your completed healthy self-care activities from the previous day. You will also have a short weekly questionnaire to complete asking about your overall mood for that week.

If you are in the passive condition, you will have a short weekly questionnaire to complete asking about your overall mood for that week.

# Permission to Take Part in a Human Research Study

At the end of the month, regardless of your condition assignment, you will complete a follow-up survey. For taking part in this study, you will receive \$20 for completing the initial questionnaire, and \$20 for the one-month follow-up questionnaire, as well as an additional \$30 for completing 90% or more of your daily checklists (a total of 25) for your time and effort if you are randomized to the enjoyable activities or healthy self-care behaviors conditions. Payment will be in the form of digital gift cards (i.e., Amazon gift card).

### What are my responsibilities if I take part in this research?

If you take part in this research, you will be responsible for: completing at least two enjoyable/healthy behaviors everyday for the next four weeks (depending on group assignment), completing short daily checklist regarding enjoyable/healthy behaviors for the next four weeks (depending on group assignment), completing short weekly surveys over the next four weeks (all group assignments), and completing pre- and post-intervention surveys (all group assignments).

# What happens if I say yes, but I change my mind later?

You can leave the research at any time it will not be held against you.

# Is there any way being in this study could be bad for me? (Detailed Risks)

Participation in this study will require describing your thoughts and behaviors, which may be uncomfortable for you. Any sensitive or personal information revealed throughout participation in this study will be stored separately from identifiable information in order to protect your privacy. Because this is a research study, there may be additional risks that we cannot identify at this time.

# What happens to the information collected for the research?

Efforts will be made to limit the use and disclosure of your personal information, including research study and medical records, to people who have a need to review this information. We cannot promise complete secrecy. Organizations that may inspect and copy your information include the IRB and other representatives of this organization.

If identifiers are removed from your identifiable private information or identifiable samples that are collected during this research, that information or those samples could be used for future research studies or distributed to another investigator for future research studies without your additional informed consent.

#### What else do I need to know?

If you agree to take part in this research study, we will pay you \$20 for completing the initial survey, and \$20 for the follow-up survey, as well as an additional \$30 for completing 90% or more of your daily checklists (a total of 25) for your time and effort depending on group assignment (i.e., enjoyable activities or healthy self-care behaviors conditions). Payment will be in the form of digital gift cards (i.e., Amazon gift card). This study will be conducted completely online.

#### MOD00003127 FSU IRB Approved 8 February 2023 

# Permission to Take Part in a Human Research Study

# **Signature Block for Capable Adult**

Your signature documents your permission to take part in this research.

| Signature of subject | Date |
|------------------------------------------|------|
| Printed name of subject | |
| Signature of person obtaining consent | Date |
| Printed name of person obtaining consent | |